CLINICAL TRIAL: NCT05730218
Title: A Phase 2, Randomized, Sham-Controlled, Single-Masked, Dose-Ranging, Multi-Center Study to Assess the Safety and Efficacy of Intravitreal ONL1204 Ophthalmic Solution in Subjects With Macula-off Rhegmatogenous Retinal Detachment
Brief Title: A Phase 2 Study to Assess the Safety and Efficacy of Intravitreal ONL1204 Ophthalmic Solution in Subjects With Mac-off Retinal Detachment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ONL Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ONL1204-RRD-002
Record Dates: First submitted 2023-02-07; First posted 2023-02-15 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Rhegmatogenous Retinal Detachment - Macula Off

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Treatment Group A (Experimental): ONL1204 Ophthalmic Solution Dose A administered by intravitreal injection
  Interventions: Drug: ONL1204 Ophthalmic Solution
- Treatment Group B (Experimental): ONL1204 Ophthalmic Solution Dose B administered by intravitreal injection
  Interventions: Drug: ONL1204 Ophthalmic Solution
- Treatment Group C (Sham Comparator): Sham injection is performed by touching the eye surface with a syringe without a needle
  Interventions: Drug: Sham treatment

INTERVENTIONS:
Drug: ONL1204 Ophthalmic Solution — ONL1204 Ophthalmic Solution at one of two doses delivered via intravitreal injection
  Arms: Treatment Group A; Treatment Group B
Drug: Sham treatment — Sham injection is performed by touching the eye surface with a syringe without a needle
  Arms: Treatment Group C

SUMMARY:
The goal of this Phase 2 clinical trial is to learn about ONL1204 Ophthalmic Solution in terms of safety and how well the drug works in patients that have a macula-off (central point of vision) rhegmatogenous retinal detachment (RRD). The main questions it aims to answer are:

* Does ONL1204 improve vision in macula-off RRD patients when used before retinal detachment repair surgery compared to patients that have surgery alone?
* Is ONL1204 safe to use as an add-on drug before retinal repair surgery?

Researchers will observe patients that receive two different dosages of ONL1204 Ophthalmic Solution (50 µg or 200 µg) compared to current standard therapy (no treatment) to see if there are differences in vision and safety outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Adult subject, ≥18 years old at the time of informed consent
2. Able and willing to give informed consent and comply with all study visits and procedures
3. Presentation with macula-off RRD with a duration ≥24 hours up to 14 days from time of central visual decline to the Baseline (Visit 2) visit, inclusive (based on subject reported date of loss of central vision) in the Study Eye (SE)
4. Visual acuity with subject's current corrective lenses or pinhole of 20/100 (line scoring) on the Snellen or ETDRS chart to light perception (LP) in the SE
5. Visual acuity with subject's current corrective lenses or pinhole of 20/200 (line scoring) or better in the fellow eye
6. Determination by Investigator of macula-off status by clinical examination with confirmation by SD-OCT or B-scan ultrasound, if available.
7. SOC retinal reattachment surgery by means of a pars plana vitrectomy (with or without scleral buckle) is indicated
8. In the opinion of the Investigator, can safely undergo the IVT injection procedure at Baseline (Visit 2)
9. Surgical repair scheduled or anticipated to take place >12 hours after IVT injection or sham (Visit 2) and ≤10 days from Screening (Visit 1)

Exclusion Criteria:

1. Presence of a complex retinal detachment (RD) in the SE, identified by one or more of the following:

   1. Giant retinal tear, defined as retinal break ≥3 clock hours in extent
   2. Proliferative vitreoretinopathy grade C1 or worse on the Retina Society Terminology Committee Classification System
   3. Presence of tractional detachments as seen in proliferative retinopathies
   4. RRD in the setting of open- or closed-globe trauma
   5. RRD following endophthalmitis or infectious retinitis
   6. Similarly complex RD as determined by the Investigator
2. Use of silicone oil tamponade in the primary RD repair without planned removal by end of study
3. Vitreous hemorrhage or cataract in the SE that prohibits adequate examination for other exclusion criteria, per Investigator's discretion
4. Presence of ocular or periocular infection or intraocular inflammation in either eye
5. Uncontrolled glaucoma, as defined by an IOP >36 mmHg in either eye, at Screening
6. Any other significant ocular disease in the SE that, in the opinion of the Investigator, would preclude a postoperative (post-op) visual acuity of at least 20/30
7. History of previous ocular surgery in the SE for RD (excluding only barrier laser), endophthalmitis, glaucoma tube shunts, trabeculectomy, or ocular trauma
8. Any systemic condition or ocular condition in either eye that, in the opinion of the Investigator, makes the subject unsuitable for treatment with an investigational agent or that would compromise the safety and tolerability of assessments in the trial
9. History of and/or active:

   1. Autoimmune disease in active flare (i.e., not well controlled on current medications) with ocular involvement that, in the opinion of the Investigator, would impact ability to participate in the trial and/or alter the outcome of retinal reattachment surgery
   2. Ocular malignancy
   3. Proliferative diabetic retinopathy or diabetic macular edema or uveitis
10. Currently participating in other clinical trials or use of any other investigational drugs or devices within 12 weeks prior to Visit 1
11. Females who are pregnant or lactating, and women of childbearing potential (WOCBP) or men with female partners of childbearing potential who are not using at least one adequate contraceptive precaution (e.g., intrauterine device, oral contraceptive, barrier method, or other contraception deemed adequate by the Investigator)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2023-04-04 (Actual); Primary Completion 2024-02-21 (Actual); Study Completion 2024-02-21 (Actual)

PRIMARY OUTCOMES:
Mean area under the log contrast sensitivity function (AULCSF) | Week 24
  Mean AULCSF as measured with the Adaptive Sensory Technology (AST) Manifold Contrast Vision Meter at Week 24 for subjects who do not have primary surgical failure.

SECONDARY OUTCOMES:
AULCSF | Week 12
Mean best-corrected visual acuity (BCVA) measured in logarithm of the minimum angle of resolution (logMAR) | Week 12
BCVA | Week 24

CONTACTS AND LOCATIONS:
Locations (36):
- United States (36):
  - Associated Retina Consultants, Phoenix, Arizona
  - Retina Associates SW PC, Tucson, Arizona
  - Win Retina, Arcadia, California
  - Global Research Management, Inc., Glendale, California
  - Salehi Retina Institute, Inc., Huntington Beach, California
  - Florida Retina Institute, Jacksonville, Florida
  - Florida Retina Consultants, Lakeland, Florida
  - Retina Specialty Institute, Pensacola, Florida
  - Sarasota Retina Institute, Sarasota, Florida
  - Retina Vitreous Associates of Florida, St. Petersburg, Florida
  - Retina Specialists of Tampa, Wesley Chapel, Florida
  - Marietta Eye Clinic, Marietta, Georgia
  - Retina Associates, Ltd., Elmhurst, Illinois
  - Retina Associates, Ltd, Elmhurst, Illinois
  - Midwest Eye Institute, Carmel, Indiana
  - Cumberland Valley Retina Consultants, Hagerstown, Maryland
  - University of Michigan Kellogg Eye Center, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - The Retina Institute, St Louis, Missouri
  - Retina Vitreous Surgeons of CNY, PC, Liverpool, New York
  - Retina Associates of Western NY, PC, Rochester, New York
  - Velocity Clinical Research, Inc., Cincinnati, Ohio
  - Oregon Health & Science University - Casey Eye Institute, Portland, Oregon
  - Erie Retina Research, LLC, Erie, Pennsylvania
  - Charleston Neuroscience Institute, Ladson, South Carolina
  - Palmetto Retina Center, LLC, West Columbia, South Carolina
  - Opthalmology Ltd, Sioux Falls, South Dakota
  - Southeastern Retina Associates, Chattanooga, Tennessee
  - Charles Retina Institute, Germantown, Tennessee
  - Retina Research Institute of Texas, Abilene, Texas
  - Austin Research Center for Retina, Austin, Texas
  - Retina Consultants of Texas, Beaumont, Texas
  - Valley Retina Institute, P.A., McAllen, Texas
  - San Antonio Eye Center, San Antonio, Texas
  - Retina Consultants of Texas, The Woodlands, Texas
  - Retina Center NW, PLLC, Silverdale, Washington